CLINICAL TRIAL: NCT04825041
Title: Efficacy of Hysteroscopic Bubble Test, Flow Test, and Peristalsis Test.
Brief Title: Efficacy of Hysteroscopic Bubble Test, Flow Test and Peristalsis Test.
Status: Completed | Type: Observational
Sponsor: Woman's Health University Hospital, Egypt (Other)
Responsible Party: Principal Investigator, Professor Atef Darwish, Professor of Obstetrics and Gynecology, Woman's Health University Hospital, Egypt
Other Study IDs: 2021
Record Dates: First submitted 2021-03-27; First posted 2021-04-01 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: Tubal Patency
Keywords: hysteroscopy; bubble flow test; Flow test; Peristalsis; Darwishscope
MeSH Terms: interventions — Fallopian Tube Patency Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Infertilite women: Subjected to three successive hysteroscopic tests
  Interventions: Diagnostic Test: Patency test

INTERVENTIONS:
Diagnostic Test: Patency test — Successive flow test, bubble flow test and peristalsis test

SUMMARY:
Fallopian tube (FT) function is complex. One of the main functions is transport of sperms for fertilization and transport of the embry for implantation. Hysteroscopic access to "Darwish Hysteroscopic Triad" allows excellent way to assess FT patency. This study compares three ways of assessing FT patency separably or in combination: flow test, bubble flow test and peristalsis test. Combined bubble flow test and peristalsis test is recently published and coined (Darwishscope)1.

DETAILED DESCRIPTION:
This study includes infertile women subjected to combined hysteroscopy and laparoscopy UGA. During hysteroscopy, on each side, three patency test are done successively: flow test, bubble flow test and peristalsis test. Gold standard diagnosis of tubal patency and status is concomitant laparoscopy.

ELIGIBILITY:
Inclusion Criteria:

* infertile women
* Probably patent FT as proved by a previous hysterosalpingography or laparoscopy.
* Office setting.
* Postmenstrual
* Non use of hormones or hormonal contraceptives.

Exclusion Criteria:

Premenstrual period. Pathologic FT.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Infertility women
Sampling Method: Probability Sample
Enrollment: 155 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-09-22 (Actual); Study Completion 2022-09-27 (Actual)

PRIMARY OUTCOMES:
FT patency | 6 months
  Success of each diagnostic test to assess FT patency.

CONTACTS AND LOCATIONS:
Locations (1):
- Woman's Health University Hospital, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No